CLINICAL TRIAL: NCT03480477
Title: Adverse Childhood Experiences in Urogynecologic Patients
Acronym: ACE-UP
Status: Terminated | Type: Observational
Why Stopped: PI confirmed that this not a Clinical trial and was inadvertently entered in the system
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Yuko Komesu, Associate Professor Obstetrics & Gynecology, University of New Mexico
Other Study IDs: 18-010
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Pelvic Floor Disorders; Interstitial Cystitis; Urinary Incontinence
Keywords: Adverse Childhood Experiences
MeSH Terms: conditions — Pelvic Floor Disorders; Cystitis, Interstitial; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pelvic Floor Disorders Group: Will collect patient information from new patients who present to the Urogynecology Clinic
  Interventions: Other: ACE questionnaire
- Control Group: Will collect patient information from patients who present to Gynecologic Clinic for their annual examination
  Interventions: Other: ACE questionnaire
- Chronic Pelvic Pain Group: Will collect patient information from patients who present to their Chronic Pelvic Pain Clinic appointment
  Interventions: Other: ACE questionnaire

INTERVENTIONS:
Other: ACE questionnaire — No intervention is performed, patients will complete BRFSS Adverse Childhood experiences questionnaire

SUMMARY:
Adverse Childhood Experiences (ACEs) have been associated with negative health outcomes, yet scant information exists regarding the relationship between ACEs, Pelvic floor disorders, and Chronic Pelvic Pain. Pelvic floor disorders (dysfunction of pelvic floor structures) are increasingly common in women, negatively affect their quality of life, and certain of these are refractory to treatment. Despite scattered reports suggesting an association between childhood abuse and specific pelvic floor disorders, the overall association between ACEs & the spectrum of pelvic floor disorders is unknown. The investigators' previous work suggests that ACEs may be associated with urgency incontinence and work by others suggest ACEs may be associated with Interstitial Cystitis/Bladder Pain Syndrome. These reports are few in number and comprehensive evaluations of ACEs relative to pelvic floor disorders are lacking. The investigators long-term objective is to investigate the relationship between ACEs in patients in the Urogynecologic and Chronic Pelvic Pain population by understanding the contributions to the development of their symptomatology. The current Urogynecology study's Primary Aims are to--1a) Describe the overall prevalence of ACEs, frequency and type of ACEs in a population of women with pelvic floor disorders 1b) Describe differences in ACE prevalence compared to the general population. Secondary Aims are to-2a) Describe ACE types/domains of controls relative to specific pelvic floor diagnoses 2b) Describe their relationship with pelvic floor disorder symptom severity. The investigators central hypothesis is that ACEs are common in women with pelvic floor disorders, that ACE frequency varies by pelvic floor diagnoses, and that ACEs may have profound effects on adult women's quality of life and responsiveness to treatment. The Chronic Pelvic Pain aims, are to 1a) describe the prevalence of ACEs in women with chronic pelvic pain. 1b) To compare the prevalence of ACEs in chronic pain patients to controls. Secondary aims are to 2a) compare the frequency and ACE type/domain of controls relative to chronic pelvic pain patients. 2b) Describe their relationship to depression/anxiety and symptom severity.The positive outcome of this prospective, cross-sectional cohort study will be its description of ACE prevalence in women with pelvic floor disorders and Chronic Pelvic Pain.

DETAILED DESCRIPTION:
Adverse Childhood Experiences (ACEs) are categorized into groups of abuse, neglect, and family/household challenges. This includes psychological, physical or sexual abuse; violence against mother, living with household members who were substance abusers, mentally ill or suicidal, or imprisoned have been shown to impact long term health in adulthood. Patients with a history of ACEs are known to be at increased risk of psychological and medical complications including depression, anxiety, low self-esteem and shame, suicidal thoughts. Medical health-related risks include obesity, chronic pain, fibromyalgia,and diabetes. The Prevalence of ACEs has been evaluated in the general population, however the prevalence in the Urogynecologic and Chronic Pelvic Pain Population have never been explored.

The Urogynecologic and Chronic Pelvic Pain population is a unique population of patients that warrants exploration. It is well known that stress levels, anxiety, and depression are further increased in patient's with Urgency Urinary Incontinence (UUI )(urinary incontinence often times associated with urinary urgency, frequency or nocturia) and overactive bladder (OAB) (urinary urgency, frequency with or without incontinence) patients with a childhood history of trauma. The investigators long-term goal is to improve treatment in the Urogynecologic and Chronic Pelvic Pain population by understanding the contributions to the development of their symptomatology. Understanding childhood experiences can help determine the challenges and development of symptoms such as OAB or Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS) (pain attributed to the bladder in the absence of organic causes such as infection, present for 6 weeks) as well as the other Urogynecologic conditions, including urinary incontinence or pelvic organ prolapse.

A key gap in the literature is how childhood experiences such as abuse may be related to Urogynecologic symptoms such as OAB or Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) as well as Chronic Pelvic Pain.

The objective of this research is to describe the prevalence of Adverse Childhood Experience (ACES) in patients in the Urogynecologic and Chronic Pelvic Pain population as well as relative to the control group. The central hypothesis is that women with Interstitial Cystitis and/or OAB as well as Chronic Pelvic Pain will report higher amount of childhood exposures than the control group.

The investigators will test the central hypothesis with the following specific Urogynecologic aims:

Aim #1: To describe the prevalence of ACEs, frequency and type of childhood exposures overall in a population of women with pelvic floor disorders, as well as differences in prevalence in a control group. Hypothesis: 1a. ACE history, based on the BRFSS-ACE Module, will be prevalent in women with pelvic floor disorders and 1b. Specific pelvic floor diagnoses (OAB/UUI +/or IC/Bladder Pain) will more commonly be associated with increased ACEs than the control group.

Aim #2: To describe frequency and ACE types/domains relative to pelvic floor diagnoses (pelvic organ prolapse, stress urinary incontinence, overactive bladder and Interstitial Cystitis/Bladder Pain Syndrome) and in the control group. And to describe their relationship with depression/anxiety and symptom severity based on validated questionnaires. Hypothesis 2a: Women with OAB and/or IC/BPS will more commonly report childhood abuse and will have increased numbers of specific ACE events, compared to the control group. Hypothesis 2b: Increased numbers of ACEs will be associated with increased anxiety, depression and symptom severity in these specific pelvic floor conditions.

The investigators will test the central hypothesis with the following specific Chronic Pelvic Pain aims:

Aim#1: 1a) describe the prevalence of ACEs in women with chronic pelvic pain. 1b) To compare the prevalence of ACEs in chronic pain patients to controls. Hypothesis 1: Chronic Pelvic Pain patients have a higher rate of ACEs than controls. Aim #2: 2a) compare the frequency and ACE type/domain of controls relative to chronic pelvic pain patients. 2b) Describe their relationship to depression/anxiety and symptom severity. Hypothesis #2: Chronic Pelvic Pain patients have an increase in ACEs and ACE domains controls, as well as more symptom severity in depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Evaluated in Urogynecology Clinic or Gynecology Clinic

Exclusion Criteria:

* Currently pregnant
* Incarcerated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: For the Urogynecology group, the investigators will recruit patients who present to the University of New Mexico Urogynecology clinics. For the control group, investigators will recruit patients who present to the University of New Mexico gynecology clinic for their annual examination. For the Chronic Pelvic Pain group, patients will be recruited from the University of New Mexico Chronic Pelvic Pain clinic. Participants will be offered study enrollment if they satisfy the inclusion/exclusion criteria. In general, the investigators will recruit study participants at their initial Urogynecology appointment, Chronic Pelvic Pain clinic and participants who present for their annual Gynecologic examination.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Prevalence | we will enroll patients in the study over the course of one year
  Report the overall prevalence of ACEs in women with pelvic floor disorders and chronic pelvic pain patients and compare the prevalence of ACEs to a control group

SECONDARY OUTCOMES:
Describe the frequency and ACE types/domains | we will enroll patients in the study over the course of one year
  To describe frequency & ACE types/domains relative to pelvic floor diagnoses (pelvic organ prolapse, stress urinary incontinence, overactive bladder and Interstitial Cystitis/Bladder Pain) and Chronic Pelvic Pain as well as the control group and to describe their relationship with depression/anxiety & symptom severity based on validated questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Yuko Komesu, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Clinics, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Dube SR, Anda RF, Felitti VJ, Chapman DP, Williamson DF, Giles WH. Childhood abuse, household dysfunction, and the risk of attempted suicide throughout the life span: findings from the Adverse Childhood Experiences Study. JAMA. 2001 Dec 26;286(24):3089-96. doi: 10.1001/jama.286.24.3089. PMID 11754674
- [Background] Anda RF, Felitti VJ, Bremner JD, Walker JD, Whitfield C, Perry BD, Dube SR, Giles WH. The enduring effects of abuse and related adverse experiences in childhood. A convergence of evidence from neurobiology and epidemiology. Eur Arch Psychiatry Clin Neurosci. 2006 Apr;256(3):174-86. doi: 10.1007/s00406-005-0624-4. Epub 2005 Nov 29. PMID 16311898
- [Background] Swift SE. The distribution of pelvic organ support in a population of female subjects seen for routine gynecologic health care. Am J Obstet Gynecol. 2000 Aug;183(2):277-85. doi: 10.1067/mob.2000.107583. PMID 10942459
- [Background] Hendrix SL, Clark A, Nygaard I, Aragaki A, Barnabei V, McTiernan A. Pelvic organ prolapse in the Women's Health Initiative: gravity and gravidity. Am J Obstet Gynecol. 2002 Jun;186(6):1160-6. doi: 10.1067/mob.2002.123819. PMID 12066091
- [Background] Jelovsek JE, Barber MD. Women seeking treatment for advanced pelvic organ prolapse have decreased body image and quality of life. Am J Obstet Gynecol. 2006 May;194(5):1455-61. doi: 10.1016/j.ajog.2006.01.060. PMID 16647928
- [Background] Lai HH, Rawal A, Shen B, Vetter J. The Relationship Between Anxiety and Overactive Bladder or Urinary Incontinence Symptoms in the Clinical Population. Urology. 2016 Dec;98:50-57. doi: 10.1016/j.urology.2016.07.013. Epub 2016 Jul 19. PMID 27450939
- [Background] Lai HH, Shen B, Rawal A, Vetter J. The relationship between depression and overactive bladder/urinary incontinence symptoms in the clinical OAB population. BMC Urol. 2016 Oct 6;16(1):60. doi: 10.1186/s12894-016-0179-x. PMID 27716241
- [Background] Kanter G, Volpe KA, Dunivan GC, Cichowski SB, Jeppson PC, Rogers RG, Komesu YM. Important role of physicians in addressing psychological aspects of interstitial cystitis/bladder pain syndrome (IC/BPS): a qualitative analysis. Int Urogynecol J. 2017 Feb;28(2):249-256. doi: 10.1007/s00192-016-3109-2. Epub 2016 Aug 31. PMID 27581769
- [Background] Nickel JC, Tripp DA, Pontari M, Moldwin R, Mayer R, Carr LK, Doggweiler R, Yang CC, Mishra N, Nordling J. Childhood sexual trauma in women with interstitial cystitis/bladder pain syndrome: a case control study. Can Urol Assoc J. 2011 Dec;5(6):410-5. doi: 10.5489/cuaj.11110. PMID 22154637
- [Background] Jundt K, Scheer I, Schiessl B, Pohl K, Haertl K, Peschers UM. Physical and sexual abuse in patients with overactive bladder: is there an association? Int Urogynecol J Pelvic Floor Dysfunct. 2007 Apr;18(4):449-53. doi: 10.1007/s00192-006-0173-z. Epub 2006 Aug 18. PMID 16917674
- [Background] Lai HH, Morgan CD, Vetter J, Andriole GL. Impact of childhood and recent traumatic events on the clinical presentation of overactive bladder. Neurourol Urodyn. 2016 Nov;35(8):1017-1023. doi: 10.1002/nau.22872. Epub 2015 Sep 1. PMID 26332868
- [Background] Centers for Disease Control and Prevention (CDC). Adverse childhood experiences reported by adults --- five states, 2009. MMWR Morb Mortal Wkly Rep. 2010 Dec 17;59(49):1609-13. PMID 21160456
- See also: Behavioral Risk Factor Surveillance System — http://www.cdc.gov/brfss/state_info/coordinators.htm